CLINICAL TRIAL: NCT03330704
Title: Randomized Controlled Trial for the Use of Patient Tailored Balanced Hypertonic Solutions in Patients With Cerebral Edema
Brief Title: Small-Volume, Patient-Specific, Balanced Hypertonic Fluid Protocol Validation
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: lack of eligible study participants
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Tim Angelotti, Associate Professor of Anesthesiology, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-43653
Record Dates: First submitted 2017-10-23; First posted 2017-11-06 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2019-02

CONDITIONS: Cerebral Edema; Saline Solution, Hypertonic
MeSH Terms: conditions — Brain Edema | interventions — Sodium Chloride; Sodium Bicarbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Therapy (Active Comparator): This group will receive 3% hypertonic sodium chloride for the management of their cerebral edema. 3% Sodium Chloride is the generic name of this intravenous fluid preparation.
  Interventions: Drug: 3% Sodium Chloride
- Balanced Therapy (Experimental): This group will undergo two simultaneous infusions. 23.4% sodium chloride and 8.4% sodium bicarbonate will be infused at the same time in various ratios for management of cerebral edema with a balanced approach
  Interventions: Drug: 23.4% Sodium Chloride; Drug: 8.4% Sodium Bicarbonate

INTERVENTIONS:
Drug: 3% Sodium Chloride — 3% sodium chloride will be infused into patients for the treatment or prevention of raised intracranial pressure
  Arms: Standard Therapy
Drug: 23.4% Sodium Chloride — 23.4% sodium chloride will be infused into patients for the treatment or prevention of raised intracranial pressure
  Arms: Balanced Therapy
Drug: 8.4% Sodium Bicarbonate — 8.4% sodium bicarbonate will be infused into patients for the treatment or prevention of raised intracranial pressure
  Arms: Balanced Therapy

SUMMARY:
Many patients with traumatic brain injuries (including strokes, blood clots, or other brain injuries) are given concentrated salt water solutions (hypertonic saline) in order to treat brain swelling (cerebral edema). Current therapies consist of a mixture of sodium and chloride, which can lead to high levels of serum chloride and increased total body water. High levels of chloride can cause acidosis, which can cause the body to function sub-optimally. Therefore, the investigators are proposing to use two concentrated solutions in these patients at the same time that will allow for a lower total volume of solution administration and reduce the rise in chloride to prevent acidosis. The main outcome will therefore be the patients sodium level, chloride level and serum pH.

ELIGIBILITY:
Inclusion Criteria:

* Able to consent
* 18 years or older
* English speaking
* Clinical indication (intracranial hypertension from cerebral edema) for hypertonic fluid administration

Exclusion Criteria:

* Fails to consent
* < 18 years old
* Hypertonic therapy not indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Total volume of intravenous hypertonic fluid administered to the patient | The fluid will be infused until the new serum sodium goal is achieved. This outcome measure will be assessed 1 week after study enrollment
  Total hypertonic fluid volume administered to each group of patients measured in milliliters of fluid.

SECONDARY OUTCOMES:
Urine output | Urine output during active hypertonic fluid infusion will be measured. This outcome measure will be assessed 1 week after study enrollment
  Urine output will be collected and measured quantitatively in milliliter units.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Angelotti, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Hospital, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share data

REFERENCES:
- [Background] Wilcox CS. Regulation of renal blood flow by plasma chloride. J Clin Invest. 1983 Mar;71(3):726-35. doi: 10.1172/jci110820. PMID 6826732
- [Background] Toung TJ, Nyquist P, Mirski MA. Effect of hypertonic saline concentration on cerebral and visceral organ water in an uninjured rodent model. Crit Care Med. 2008 Jan;36(1):256-61. doi: 10.1097/01.CCM.0000295306.52783.1E. PMID 18090381
- [Background] Diringer MN, Zazulia AR. Osmotic therapy: fact and fiction. Neurocrit Care. 2004;1(2):219-33. doi: 10.1385/NCC:1:2:219. PMID 16174920
- [Background] Erdman MJ, Riha H, Bode L, Chang JJ, Jones GM. Predictors of Acute Kidney Injury in Neurocritical Care Patients Receiving Continuous Hypertonic Saline. Neurohospitalist. 2017 Jan;7(1):9-14. doi: 10.1177/1941874416665744. Epub 2016 Aug 29. PMID 28042364
- [Background] Neavyn MJ, Boyer EW, Bird SB, Babu KM. Sodium acetate as a replacement for sodium bicarbonate in medical toxicology: a review. J Med Toxicol. 2013 Sep;9(3):250-4. doi: 10.1007/s13181-013-0304-0. PMID 23636658